CLINICAL TRIAL: NCT05292014
Title: ANGIOLITE Post-Market Clinical Follow-up Study
Brief Title: ANGIOLITE PMCF Study ( rEPIC04F )
Acronym: rEPIC04F
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: ANGIOLITE PMCF Study
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: ANGIOLITE

INTERVENTIONS:
Device: ANGIOLITE — Patients in whom treatment with ANGIOLITE has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Angiolite sirolimus eluting stent to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Angiolite sirolimus eluting stent.

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the Angiolite Sirolimus Eluting Stent in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with ANGIOLITE according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

• Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with ANGIOLITE according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, stent thrombosis (Academic Research Consortium definitive/ probable), and new Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom fromTarget Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).
Freedom from Accidental dislodgement of the stent | During percutaneous coronary intervention (PCI)
  Freedom from Accidental dislodgement of the stent
Freedom from Balloon rupture | During PCI
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI
  Freedom from Hypotube rupture
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - H. Puerta Del Mar, Cadiz
  - Hospital Universitario de Leon, León
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Sigwart U, Puel J, Mirkovitch V, Joffre F, Kappenberger L. Intravascular stents to prevent occlusion and restenosis after transluminal angioplasty. N Engl J Med. 1987 Mar 19;316(12):701-6. doi: 10.1056/NEJM198703193161201. PMID 2950322
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Stone GW, Moses JW, Ellis SG, Schofer J, Dawkins KD, Morice MC, Colombo A, Schampaert E, Grube E, Kirtane AJ, Cutlip DE, Fahy M, Pocock SJ, Mehran R, Leon MB. Safety and efficacy of sirolimus- and paclitaxel-eluting coronary stents. N Engl J Med. 2007 Mar 8;356(10):998-1008. doi: 10.1056/NEJMoa067193. Epub 2007 Feb 12. PMID 17296824
- [Background] Wu X, Li L, He L. Drug-Coated Balloon versus Drug-Eluting Stent in Patients with Small-Vessel Coronary Artery Disease: A Meta-Analysis of Randomized Controlled Trials. Cardiol Res Pract. 2021 Apr 13;2021:1647635. doi: 10.1155/2021/1647635. eCollection 2021. PMID 33953973